CLINICAL TRIAL: NCT01741922
Title: Effectiveness of the Timing of the Administration of Aspirin in Hypertensive Patients Treated With Low Doses of Acetyl Salicylic Acid for Secondary Prevention - TAHPS
Brief Title: Effectiveness of Night Administration of Low Dose Aspirin in Hypertensive Patients
Acronym: TAHPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Spanish Clinical Research Network - SCReN (Network); Public Health Service of Cataluña (Other)
Responsible Party: Principal Investigator, Victoria Ruiz Arzalluz, Primary Care Practitioner in Basque Health Service, Basque Health Service
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TAHPS-2011-004760-29
Record Dates: First submitted 2012-11-07; First posted 2012-12-05 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Low dose; aspirin; ASA; Hypertension; blood pressure
MeSH Terms: conditions — Hypertension | interventions — Contraceptives, Oral; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASA evening&placebo morning (Experimental): Patients will receive acetylsalicylic acid (100 mg)in the evening and placebo in the morning.
  Interventions: Drug: ASA evening; Drug: Placebos morning
- ASA morning&placebo evening (Active Comparator): Patients will receive acetylsalicylic acid (100 mg) in the morning and placebo in the evening
  Interventions: Drug: Acetylsalicylic morning; Drug: Placebo evening

INTERVENTIONS:
Drug: ASA evening — Patients will be assigned to one of two parallel groups: Active comparator group during the first two months, namely, administration of acetylsalicylic acid 100 mg, in the morning and placebo in the evening and Experimental: Acetylsalicylic acid in the evening & placebo in the morning group, of administration of acetylsalicylic acid 100 mg in the evening, between (20.00 and 22.00 hours) and placebo in the morning. After that, patients will then undergo a washout period of 15 days to one month, during which all patients participating in the study will take their ASA doses during the daytime. After the washout period, participants will exchange groups
  Other Names: ASA; Low dose; aspirine
  Arms: ASA evening&placebo morning
Drug: Acetylsalicylic morning — Patients will be assigned in a blind and randomized way to one of two parallel groups: group I with the control treatment during the first two months, namely, administration of aspirin 100 mg, in the morning and placebo in the evening and group II initially receiving the intervention, of administration of aspirin 100 mg in the evening, between (20.00 and 22.00 hours) and placebo in the morning. After that, patients will then undergo a washout period of 15 days to one month, during which all patients participating in the study will take their ASA doses during the daytime. After the washout period, participants will exchange groups, i.e., patients randomly allocated to group I, so having taken aspirin in the morning and placebo in the evening, will now receive the intervention treatment, namely, administration of ASA in the evening and placebo in the morning for another two months and vice verse.
  Other Names: Asa; Low dose; aspirine
  Arms: ASA morning&placebo evening
Drug: Placebos morning — Patients will be assigned to one of two parallel groups: Active comparator group during the first two months, namely, administration of acetylsalicylic acid 100 mg, in the morning and placebo in the evening and Experimental: Acetylsalicylic acid in the evening & placebo in the morning group, of administration of acetylsalicylic acid 100 mg in the evening, between (20.00 and 22.00 hours) and placebo in the morning. After that, patients will then undergo a washout period of 15 days to one month, during which all patients participating in the study will take their ASA doses during the daytime. After the washout period, participants will exchange groups
  Arms: ASA evening&placebo morning
Drug: Placebo evening — Patients will be assigned to one of two parallel groups: Active comparator group during the first two months, namely, administration of acetylsalicylic acid 100 mg, in the morning and placebo in the evening and Experimental: Acetylsalicylic acid in the evening & placebo in the morning group, of administration of acetylsalicylic acid 100 mg in the evening, between (20.00 and 22.00 hours) and placebo in the morning. After that, patients will then undergo a washout period of 15 days to one month, during which all patients participating in the study will take their ASA doses during the daytime. After the washout period, participants will exchange groups
  Arms: ASA morning&placebo evening

SUMMARY:
The goal is to investigate in patients with high blood pressure, BP, namely, those with systolic blood pressure and diastolic blood pressure, SBP/DBP higher than or equal to 140/90 mmHg, and high cardiovascular risk, under treatment with low-dose acetylsalicylic acid, ASA, whether changing the time they take the drug (same dose) to bedtime (from taking it at some point during the active part of the day) produces a drop in their blood pressure (mean systolic and diastolic over 24 hours) of at least 2.5 mm Hg; and also whether among non-dippers, under secondary treatment with low-dose ASA, there is be a greater decrease in their night BP when the drug is taken in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients (≥140/90)
* Patients from 18 to 80 years old
* Patients are currently taking low doses of ASA during the day, for secondary prevention of cardiovascular events
* Patients have been stable for at least one month with their current antihypertensive and antiplatelet therapy.

Exclusion Criteria:

* Severe and/or terminal illness
* Moderate/severe congestive heart failure (CHF), New York Heart Association, NYHA stage ≥ III
* Moderate/severe chronic renal failure glomerular filtration rate <45ml/min.
* Physical or mental illness that prevents the patient´s collaboration
* Being a heavy drinker, consuming more than 280 g of alcohol per week in the case of men or 170 g for women31
* Concomitant treatment with other antiplatelets or anticoagulants
* Taking nonsteroidal antiinflammatory drugs, NSAIDs, on a regular basis
* Treatment with ASA at doses outside those established in the inclusion criteria (above)
* ASA already being taken in the evening
* Being a shift worker or having a very intensive work schedule
* Hospital admission during the clinical trial
* Changes being made in the antihypertensive and antiplatelet therapy taken by the patient during the seven months of the trial
* Patients with unstable treatment or clinical condition requiring frequent adjustments thereof.
* Compliance with less than 90% of the doses, both those for daytime and those for evening administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mean SBP and DBP measured with Ambulatory Blood Pressure Monitoring (ABPM) over a 24 hour period | Change from baseline in sistolyc blood pressure at five months
  To evaluate the effect of evening administration of low doses of aspirin (100 mg) on the BP of hypertensive patients with high cardiovascular risk, comparing with the effect of day administration, we are going to measure the change in the mean SBP and DBP measured with Ambulatory Blood Pressure Monitoring (ABPM) over a 24 hour period from baseline at the end of the study, five months later.

SECONDARY OUTCOMES:
Mean of day/night SBP and DBP ratios measured with Ambulatory Blood Pressure monitoring Monitoring | Change from baseline in sistolyc blood pressure at five months
  To optimize the control of BP in hypertensive patients treated with low doses of aspirin for secondary prevention. We are going to describe the changes in day-night pattern of BP as a function of the time of administration of low doses of aspirin in non-dipper patients, objectified by the mean of day:night SBP and DBP ratios.
The mean of heart rate (HR) and the mean of pulse pressure (PP) | Change from baseline in sistolyc blood pressure at five months
  To optimize the control of BP in hypertensive patients treated with low doses of aspirin for secondary prevention. We are going to identify any changes in the mean of heart rate (HR) and the mean of pulse pressure (PP) with evening administration of ASA.
Percentage of adverse events related to ASA evening administration versus day administration | Change from baseline in sistolyc blood pressure at five months
  we are going to measured the percentage of adverse events at the end of the study to assess any changes in the side effects of aspirin when it is taken in the evening compared to day-time administration.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ruíz, Dr., Principal Investigator — Basque Health Service
Locations (3):
- Spain (3):
  - Primary Care Research Unit of Bizkaia, Bilbao, Bizkaia
  - Primary care of IDIAP Jordi Gol, Barcelona, Catalonia
  - Primary Care Research Unit of Bizkaia, Gipuzkoa Oeste, Gipuzkoa

REFERENCES:
- [Background] Ruiz-Arzalluz MV, Fernandez MC, Burgos-Alonso N, Vinyoles E, San Vicente Blanco R, Grandes G; TAHPS group. Protocol for assessing the hypotensive effect of evening administration of acetylsalicylic acid: study protocol for a randomized, cross-over controlled trial. Trials. 2013 Jul 27;14:236. doi: 10.1186/1745-6215-14-236. PMID 23890047
- [Derived] Ruiz Arzalluz MV, Burgos-Alonso N, Garcia-Alvarez A, Gomez Fernandez MC, Vinyoles E, Grandes G; TAHPS Group. Evaluation of the antihypertensive effect of nocturnal administration of acetylsalicylic acid: a cross-over randomized clinical trial. J Hypertens. 2019 Feb;37(2):406-414. doi: 10.1097/HJH.0000000000001887. PMID 30095728